CLINICAL TRIAL: NCT05097833
Title: KS, NE, and TX Fathers, Couples, and Co-parents Whose Children Are Involved in the Child Welfare System Will Gain the Skills and Knowledge to be Better Parents Through Saint Francis Fatherhood FIRE
Brief Title: Local Evaluation of the Saint Francis Ministries Fatherhood FIRE Program
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 146802
Record Dates: First submitted 2021-10-01; First posted 2021-10-28 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2024-04

CONDITIONS: Parenting; Parent-Child Relations; Relationship, Marital; Relationship, Family; Relationships, Father-Child; Fathers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Treatment Group (Experimental): Randomized group of participants receiving an enhanced Fatherhood FIRE program.
  Interventions: Behavioral: Enhanced Saint Francis Fatherhood FIRE Program
- Control Group (Active Comparator): Randomized group of participants receiving the 'services as usual' Fatherhood program.
  Interventions: Behavioral: Services as Usual Saint Francis Fatherhood FIRE Program

INTERVENTIONS:
Behavioral: Enhanced Saint Francis Fatherhood FIRE Program — Fathers receive an enhanced series of pro-parenting, relationship, and economic stability workshops over 16 weeks. Workshop series are based on a diverse curricula including a combination of either 24/7 Dad or Parent Project and Connections to Success and the Nurturing Fathers enhancement program.
  Arms: Enhanced Treatment Group
Behavioral: Services as Usual Saint Francis Fatherhood FIRE Program — Fathers receive the services as usual approach which includes a series of pro-parenting, relationship, and economic stability workshops over 13 weeks. Workshop series are based on a diverse curricula including a combination of either 24/7 Dad or Parent Project and Connections to Success.
  Arms: Control Group

SUMMARY:
This study is the local process and impact evaluation for Saint Francis Ministries' Fatherhood FIRE Program.

DETAILED DESCRIPTION:
This project is based on federal legislation that requires evaluation of a program being implemented and delivered by Saint Francis Ministries, a community-based non-profit organization serving children and families. Saint Francis Ministries received federal funds to expand and deliver the Fatherhood FIRE Program to community-based and justice-system involved fathers in their service area. The FIRE program, which stands for Family-Oriented, Interconnected, Resilient, and Essential, aims to promote responsible and positive fatherhood parenting practices and develop and maintain healthy relationships with their partners and other co-parents (e.g., mothers of their children). Evaluation of the program is a condition of Saint Francis Ministries' grant award from the U.S. Department of Health and Human Services. The KU evaluation team at the School of Social Welfare has been contracted by Saint Francis Ministries to conduct the evaluation. The evaluation will be carried out in two parts: 1) a process evaluation and 2 an outcomes evaluation. The process and target populations for both the process and outcomes components are as follows. PROCESS EVALUATION: The process study involves individuals involved in the implementation of the Fatherhood FIRE program at Saint Francis Ministries. Specific populations eligible for inclusion in the process evaluation include: (1) implementation teams facilitating the Fatherhood FIRE program in three states in Saint Francis Ministries service area (Kansas, Nebraska, & Texas), (2) members of the Fatherhood FIRE Data, Assessment, and Dissemination Workgroup, an advisory group comprised of Saint Francis program administrators and the evaluation team charged with planning and overseeing data collection, evaluation, and dissemination efforts, and (3) the evaluation study team. OUTCOMES EVALUATION: Fathers ages 18 and older who are not incarcerated and are enrolled and participating in the Fatherhood FIRE program. To be eligible for inclusion in the evaluation study, program participants must not be incarcerated, have children up to age 24, and may be living with or apart from their children. Eligible participants may be biological parents, adoptive or foster parents, or other caregivers in the parenting role if they have children who meet the age criteria.

ELIGIBILITY:
Inclusion Criteria:

* Fathers with children up to 24 year old
* Fathers participating in the Saint Francis Fatherhood FIRE Program

Exclusion Criteria:

* Fathers who are incarcerated

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Intervention and evaluation is designed for fathers (males) 18 and older with children up to 24 years of age.
Enrollment: 600 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Healthy relationship and marriage skills | Measurement of the outcome will occur at three-time points: 1) Pre intervention, 2) at program completion an average of 16 weeks after pre-intervention measure, 3) 3-months post program completion
  Dads in the enhanced group demonstrate larger and more sustained change in healthy relationship and marriage skills (e.g., compromise and interactional reactivity) than the control group. The measurement tool used to assess this outcome is the Romantic Partner Conflict Scale (Zacchilli, Hendrick, & Hendrick, 2009).
Parenting skills | Measurement of the outcome will occur at three-time points: 1) Pre intervention, 2) at program completion an average of 16 weeks after pre-intervention measure, 3) 3-months post program completion
  Dads in the enhanced group demonstrate larger and more sustained change in parenting skills than the control group. The measurement tool used to assess this outcome is the Parenting Sense of Competence Scale (Ohan, Leung, & Jonston, 2000; Johnston & Mash, 1989; Gillmore & Cuskelly, 2008).
Co-parenting skills | Measurement of the outcome will occur at three-time points: 1) Pre intervention, 2) at program completion an average of 16 weeks after pre-intervention measure, 3) 3-months post program completion
  Dads in the enhanced group demonstrate larger and more sustained change in co-parenting skills than the control group. The measurement tool used to assess this outcome is the Daily Co-Parenting Scale (D-COP; McDaniel, Teti, & Feinberg, 2017).
Father-child engagement | Measurement of the outcome will occur at three-time points: 1) Pre intervention, 2) at program completion an average of 16 weeks after pre-intervention measure, 3) 3-months post program completion
  Dads in the enhanced group demonstrate larger and more sustained change in father/child engagement than the control group. The measurement tool used to assess this outcome is the Inventory of Father Involvement (Hawkins, Bradford, Palkovitz, & Christiansen, 1999).

CONTACTS AND LOCATIONS:
Overall Officials: Jared L Barton, PhD, Principal Investigator — University of Kansas
Locations (1):
- University of Kansas School of Social Welfare, Lawrence, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be archived at the end of the study through an accessible archiving site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will become available at the end of the study anticipated September 2025